CLINICAL TRIAL: NCT02452944
Title: Comparison of Nerve Stimulating Approach and Interfascial Injection Approach During Sono-guided Obturator Nerve Block in Transurethral Resection of Bladder Tumors Under Spinal Anesthesia
Brief Title: Comparison of Nerve Stimulating Approach and Interfascial Injection Approach During Sono-guided Obturator Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Mi Geum Lee, assistant professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: GAIRB2014-337
Record Dates: First submitted 2015-05-07; First posted 2015-05-25 (Estimated); Results first posted 2015-07-23 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Bladder Cancer
Keywords: nerve stimulator, obturator nerve, ultrasound
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- US-IFI group (Experimental): ultrasound-guided obturator nerve block with interfascial injection approach group (US-IFI; experimental group)
  The stimulating needle without nerve stimulator advanced via an ultrasound to position the needle tip on the fascia between adductor longus and adductor brevis muscles. 10mL of local anesthetics were slowly injected. The needle was reinserted to position the needle tip on the fascia between adductor brevis and adductor magnus muscles, another 5mL of LA was injected.
  After that, the needle was reinserted to the same spots attached with nerve stimulator at 1.0 mA. If adductor muscle twitching was shown, another 5mL of LA was injected, and it was documented as 'fail'.
  Interventions: Device: nerve stimulator (stimuplex HNS12); Device: ultrasound
- US-NS group (Active Comparator): ultrasound-guided obturator nerve block with nerve stimulating approach group (US-NS; control group) The stimulating needle attached to a nerve stimulator advanced via an ultrasound to position the needle tip on the fascia between adductor longus and adductor brevis muscles. The nerve stimulator was then turned on, and the stimulation current started at 0.5 mA. If adductor muscle twitching was observed on the sonogram even at the stimulation current 0.3mA, 10mL of local anesthetics were slowly injected. The needle was reinserted to position the needle tip on the fascia between adductor brevis and adductor magnus muscles. The stimulation current started at 0.5 mA. If adductor muscle twitching was visualized on the sonogram even at 0.3mA, another 5mL of LA was injected.
  Interventions: Device: nerve stimulator (stimuplex HNS12); Device: ultrasound

INTERVENTIONS:
Device: nerve stimulator (stimuplex HNS12) — whether using the nerve stimulator or not when the investigators do the ultrasound-guided obturator nerve block
Device: ultrasound — we did obturator nerve block with ultrasound guided method for searching the fascias where the anterior and posterior branches of obturator nerve run.

SUMMARY:
Transurethral resection of bladder tumor (TURB) has been essential treatment for bladder tumours. Direct electrical stimulation of an obturator nerve during the TURB procedures can trigger an inadvertent adductor muscle spasm, which can cause a serious complication like bladder perforation.

General anesthesia with muscle relaxants for TURB does not guarantee a prevention of the adductor muscle spasm. Spinal anesthesia with selective obturator nerve block (ONB) can be an alternative anesthesia for TURB, but adductor spasm can also be induced because of incomplete ONB. Recently, ultrasound guidance with nerve stimulator has been used to enhance the safety, efficacy and shortening the onset time of ONB.

Some papers describe that comparable ONB can be done using ultrasound only without nerve stimulator, in which there is a principle that obturator nerve runs along a given pathway. Basically, obturator nerve is divided into two branches after exiting the obturator canal. The anterior branch is located in the fascial planes among adductor longus, adductor brevis and pectineus muscles, and the posterior branch is located between the adductor brevis and adductor magnus muscles at the inguinal area. But it has been known that there are many branching patterns of obturator nerve and high anatomic variability in the inguinal area in a cadaver study. And subdivisions of obturator nerve in the inguinal area have been described.

Therefore, this study was conducted to investigate the success rate of ultrasound-guided obturator nerve block with interfascial injection approach group (US-IFI; experimental group) was comparable to ultrasound-guided obturator nerve block with nerve stimulating approach group (US-NS; control group) in TURB under spinal anesthesia. And we also evaluated adductor muscle twitching patterns at the inguinal region when the ONB was performed.

DETAILED DESCRIPTION:
After obtaining approval from the Gachon Gil Hospital Ethical Committee, written informed consent was obtained from all patients anticipating TURB with American Society of Anesthesiologists physical status (ASA) I or II. Sixty two patients anticipating transurethral resection of the bladder tumors (TURB) under spinal anesthesia were enrolled in this randomized controlled trial from December 2014 to May 2015. Exclusion criteria included patients with diabetes or peripheral neuropathy; motor or sensory deficits in the lower extremities, ASA greater than III, coagulation disorders, anticoagulant medication, known allergy to local anesthetics, contraindications for spinal anesthesia (infection at injection site, severe scoliosis or fusion operation), uncooperative patients and patients' refusal. Routine monitoring was begun and Spinal anesthesia with hyperbaric 0.5% bupivacaine 12-15 mg was performed to reach the level of anesthesia, at least T10 to T4 in all patients.

Patients were then randomized into 1 of 2 groups (US-NS vs US-IFI) to receive ONB in the inguinal crease level. Randomization was performed by a computer-generated random numbers table. We counted one side obturator nerve as one, the number. Whether the right or left ONB was done, was decided by surgeon according to the tumor location. If obturator block was done in both sides, let it belong to the same group, and we counted it as two, the number.

Patients were then positioned supine, and the affected leg was slightly abducted and rotated externally without knee flexion, and the inguinal region was prepared with a povidone iodine solution. The 10 MHz linear probe (Zonare Medical Systems, California, USA) equipped with a sterile plastic cover and gel. The transducer was positioned parallel to the inguinal crease with 90° to the skin with the image depth of 4-5 cm. The inguinal region was examined laterally from the femoral vein until the 3 muscle layers consisting of the adductor longus, adductor brevis, and adductor magnus were identified with pectineus muscle medially along the inguinal crease. We allowed transducer tilting cranially 0°-20° angle until a fascial planes of the pectineus and adductor muscles were identified. A thick hyperechoic fascia was used as a targeting landmark for ONB, not focus on the obturator nerve itself (One between adductor longus and adductor brevis muscles for anterior branch, another between adductor brevis and adductor magnus muscles for posterior branch of obturator nerve). We excluded the case, in which three muscle layers were not identified definitely within the range.

In the US-NS group, 22-gauge, 120-mm stimulating needle (Stimuplex insulated needle; D Plus B. Braun, Melsungen, Germany) attached to a nerve stimulator (Stimuplex HNS12;B. Braun, Melsungen, Germany) advanced via an ultrasound in-plane approach from lateral to medical direction to position the needle tip on the anterior branch. The nerve stimulator was then turned on, and the stimulation current started at 0.5 mA. If adductor muscle twitching was observed on the sonogram even at the stimulation current 0.3mA, 10mL of local anesthetics (LA; 1.5% lidocaine + epi 1:200,000) were slowly injected within the muscle interface after negative aspiration, resulting in separation of these two muscles under real-time visualization. If there was misdistribution of LA spread (eg, spread into the muscle tissue), the needle was redirected until the correct spread of LA was visualized. The needle was withdrawn to the skin and reinserted to position the needle tip on the posterior branch. The stimulation current started at 0.5 mA. If adductor muscle twitching was visualized on the sonogram even at 0.3mA, another 5mL of LA was injected. After injection to the anterior and posterior branch, the stimulation current increased 1.0 mA, and needle was re-advanced as like Fig 1d for searching the residual muscle twitching. If muscle twitching was observed, then current was decreased to 0.5 mA, and confirming the muscle twitching on the sonogram at that current, 5ml of LA injected. We wrote that muscle twitching was occurred in what kind of muscles or fascias.

In the US-IFI group, 22-gauge, 120-mm stimulating needle (Stimuplex insulated needle; D Plus B. Braun, Melsungen, Germany) without nerve stimulator advanced via an ultrasound in-plane approach from lateral to medical direction to position the needle tip on anterior branch. After negative aspiration, 10mL of LA were slowly injected within the muscle interface, resulting in separation of these two muscles under real-time visualization. The needle was withdrawn to the skin and reinserted to position the needle tip on posterior branch, another 5mL of LA was injected. After that, the needle was withdrawn to the skin and reinserted to the same spots, attached with nerve stimulator at the stimulation current 1.0 mA for confirming the block of anterior and posterior branch. If adductor muscle twitching was shown on sonogram, another 5mL of LA was injected, and it was documented as 'fail'. After that, needle was re-advanced as like US-NS group for searching the residual muscle twitching. It then went through the same process as the US-NS group, and we wrote that muscle twitching was occurred in what kind of muscles or fascias. We used only the nerve stimulator for confirming the success or fail of the ONB before the TURB surgery.

Any needle redirection after withdrawing to the skin, was recorded as an additional needle pass. Before the injection, the image was captured as static, and the depth of anterior and posterior branch was measured by use of the built-in caliper of the ultrasound machine. We recorded ONB time, and time from the start of the sonographic examination until muscle layers identification was included. All blocks were performed by one anesthesiologist with more than 60 ONB experiences.

After performing the ONB, patients were positioned in lithotomy position. Endoscopic resection of the neoplasm was started using a bipolar resectoscope (electrical current: 280 W) and endovesical irrigation with a normal saline solution. The surgery was performed by six surgeons randomly. We requested two assistants of urology, who didn't know the study groups (US-NS vs US-IFI) for obturator reflex grading. Obturator reflex grade was assessed by the scale of Lee's paper. Gr I: no movement or palpable muscle twitching, Gr II: palpable muscle twitching without movement, Gr III: slight movement of the thigh not interfering with the surgical procedure, and Gr IV: vigorous movement interfering with the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* all patients anticipating transurethral resection of bladder tumors with American Society of Anesthesiologists physical status(ASA) I or II

Exclusion Criteria:

* patients with diabetes or peripheral neuropathy; motor or sensory deficits in the lower extremities, ASA greater than III, coagulation disorders, anticoagulant medication, known allergy to local anesthetics, contraindications for spinal anesthesia (infection at injection site, severe scoliosis or fusion operation), uncooperative patients and patients' refusal

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-12; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mi Geum Lee, MD, PhD, Study Director — Gachon University Gil Medical Center

REFERENCES:
- [Background] Anagnostopoulou S, Kostopanagiotou G, Paraskeuopoulos T, Chantzi C, Lolis E, Saranteas T. Anatomic variations of the obturator nerve in the inguinal region: implications in conventional and ultrasound regional anesthesia techniques. Reg Anesth Pain Med. 2009 Jan-Feb;34(1):33-9. doi: 10.1097/AAP.0b013e3181933b51. PMID 19258986

RESULTS

PARTICIPANT FLOW:
Recruitment Details: dates of the recruitment period: January 2015 - May 2015 types of location: in the operating room
Groups:
- US-IFI Group: ultrasound-guided obturator nerve block with interfascial injection approach group (US-IFI; experimental group)
  The stimulating needle without nerve stimulator advanced via an ultrasound to position the needle tip on the fascia between adductor longus and brevis muscles. 10mL of local anesthetics (LA; 1.5% lidocaine + epi 1:200,000) were injected. The needle was reinserted to position the needle tip on the fascia between adductor brevis and magnus muscles, another 5mL of LA was injected.
  After that, the needle was reinserted to the same spots attached with nerve stimulator for confirming the block. If adductor muscle twitching was shown, another 5mL of LA was injected, and it was documented as 'fail'.
- US-NS Group: ultrasound-guided obturator nerve block with nerve stimulating approach group (US-NS; control group)
  The stimulating needle attached to a nerve stimulator advanced via an ultrasound to position the needle tip on the fascia between adductor longus and brevis. The nerve stimulator was then turned on, and the stimulation current started at 0.5 mA. If adductor muscle twitching was observed on the sonogram even at the stimulation current 0.3mA, 10mL of local anesthetics (LA;1.5% lidocaine + epi 1:200,000) were slowly injected. The needle was reinserted to position the needle tip on the fascia between adductor brevis and magnus. The stimulation current started at 0.5 mA. If adductor muscle twitching was visualized on the sonogram even at 0.3mA, another 5mL of LA was injected.
Period: Overall Study
Arm/Group | US-IFI Group | US-NS Group
Started | 31 | 31
Completed | 31 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- US-IFI Group: ultrasound-guided obturator nerve block with interfascial injection approach group (US-IFI; experimental group)
  The stimulating needle without nerve stimulator advanced via an ultrasound to position the needle tip on the fascia between adductor longus and brevis. 10mL of local anesthetics were slowly injected. The needle was reinserted to position the needle tip on the fascia between adductor brevis and magnus, another 5mL of LA was injected.
  After that, the needle was reinserted to the same spots attached with nerve stimulator at 1.0 mA. If adductor muscle twitching was shown, another 5mL of LA was injected, and it was documented as 'fail'.
- US-NS Group: ultrasound-guided obturator nerve block with nerve stimulating approach group (US-NS; control group) The stimulating needle attached to a nerve stimulator advanced via an ultrasound to position the needle tip on the fascia between adductor longus and brevis. The nerve stimulator was then turned on, and the stimulation current started at 0.5 mA. If adductor muscle twitching was observed on the sonogram even at 0.3mA, 10mL of local anesthetics was injected. The needle was reinserted to position the needle tip on the fascia between adductor brevis and magnus. The stimulation current started at 0.5 mA. If adductor muscle twitching was visualized on the sonogram even at 0.3mA, another 5mL of LA was injected.
- Total: Total of all reporting groups
Arm/Group | US-IFI Group | US-NS Group | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (14) | 70 (11) | 69.2 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 25 | 25 | 50
Height (cm) [Mean (Standard Deviation); unit: cm] | 164.1 (7.6) | 166.3 (6.3) | 165.2 (7.0)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 61.9 (11.3) | 63.1 (10.2) | 62.5 (10.7)
American Society of Anesthesiologists physical status (ASA) [Number; unit: participants] — ASA class I: a normal healthy patient ASA class II: a patient with mild systemic disease
  participants
    ASA I | 7 | 11 | 18
    ASA II | 24 | 20 | 44

OUTCOME MEASURES:

1. Primary Outcome: Success Rate of Ultrasound-guided Obturator Nerve Block With US-IFI Group and US-NS Group
Description: We used only the nerve stimulator for confirming the success or fail of the ONB before the surgery, so we assumed that the US-NS group had complete ONB in all patients.
  In US-IFI group, complete ONB was confirmed with nerve stimulator at the end of the procedure, and if the residual twitching remained, the case was considered to be a 'fail'.
Time Frame: up to 8 weeks
Measure: Number; unit: participants
Groups:
- US-IFI Group: ultrasound-guided obturator nerve block with interfascial injection approach group (US-IFI; experimental group)
  The stimulating needle without nerve stimulator advanced via an ultrasound to position the needle tip on the fascia between adductor longus and adductor brevis. 10mL of local anesthetics were slowly injected. The needle was reinserted to position the needle tip on the fascia between adductor brevis and adductor magnus muscles, another 5mL of LA was injected.
  After that, the needle was reinserted to the same spots attached with nerve stimulator at 1.0 mA. If adductor muscle twitching was shown, another 5mL of LA was injected, and it was documented as 'fail'.
  nerve stimulator (stimuplex HNS12): whether using the nerve stimulator or not when the investigators do the ultrasound-guided obturator nerve block
  ultrasound: we did obturator nerve block with ultrasound guided method for searching the fascias where the anterior and posterior branches of obturator nerv
- US-NS Group: ultrasound-guided obturator nerve block with nerve stimulating approach group (US-NS; control group) The stimulating needle attached to a nerve stimulator advanced via an ultrasound to position the needle tip on the fascia between adductor longus and adductor brevis. The nerve stimulator was then turned on, and the stimulation current started at 0.5 mA. If adductor muscle twitching was observed on the sonogram even at the stimulation current 0.3mA, 10mL of local anesthetics were slowly injected. The needle was reinserted to position the needle tip on the fascia between adductor brevis and adductor magnus muscles. The stimulation current started at 0.5 mA. If adductor muscle twitching was visualized on the sonogram even at 0.3mA, another 5mL of LA was injected.
  nerve stimulator (stimuplex HNS12): whether using the nerve stimulator or not when the investigators do the ultrasound-guided obturator nerve block
  ultrasound: we did obturator nerve block with ultrasound guided m
Arm/Group | US-IFI Group | US-NS Group
Number analyzed (Participants) | 31 | 31
participants
  success | 25 | 31
  fail | 6 | 0

2. Secondary Outcome: Count the Number of Sub-divisions of Obturator Nerve at the Inguinal Crease
Description: We checked the additional intramuscular twitching with at least 3 times more needling after block the anterior and posterior branches in both groups. And documented that twitching occurred in what kind of muscles.
Time Frame: up to 8 weeks
Measure: Number; unit: participants
Groups:
- US-IFI Group: ultrasound-guided obturator nerve block with interfascial injection approach group (US-IFI; experimental group)
  The stimulating needle without nerve stimulator advanced via an ultrasound to position the needle tip on the fascia between adductor longus and brevis. 10mL of local anesthetics were slowly injected. The needle was reinserted to position the needle tip on the fascia between adductor brevis and magnus, another 5mL of LA was injected.
  After that, the needle was reinserted to the same spots attached with nerve stimulator at 1.0 mA. If adductor muscle twitching was shown, another 5mL of LA was injected, and it was documented as 'fail'.
  nerve stimulator (stimuplex HNS12): whether using the nerve stimulator or not when the investigators do the ultrasound-guided obturator nerve block
  ultrasound: we did obturator nerve block with ultrasound guided method for searching the fascias where the anterior and posterior branches of obturator nerve run.
- US-NS Group: ultrasound-guided obturator nerve block with nerve stimulating approach group (US-NS; control group) The stimulating needle attached to a nerve stimulator advanced via an ultrasound to position the needle tip on the fascia between adductor longus and brevis. The nerve stimulator was then turned on, and the stimulation current started at 0.5 mA. If adductor muscle twitching was observed on the sonogram even at 0.3mA, 10mL of local anesthetics were injected. The needle was reinserted to position the needle tip on the fascia between adductor brevis and magnus. The stimulation current started at 0.5 mA. If adductor muscle twitching was visualized on the sonogram even at 0.3mA, another 5mL of LA was injected.
Arm/Group | US-IFI Group | US-NS Group
Number analyzed (Participants) | 31 | 31
participants
  in the Adductor brevis muscle | 8 | 7
  In the adductor magnus muscle | 0 | 1
  In the Pectineus muscle | 1 | 2
  in the fascia of anterior branch run | 2 | 1
  In the fascia of posterior branch run | 2 | 4

ADVERSE EVENTS:
Time Frame: 5 months
Description: we examined the adverse events during the obturator nerve block, and reviewed the urology chart for follow-up of any neurologic or vascular complications for patient's hospitalization periods.
Groups:
- US-IFI Group: ultrasound-guided obturator nerve block with interfascial injection approach group (US-IFI; experimental group)
  The stimulating needle without nerve stimulator advanced via an ultrasound to position the needle tip on the fascia between adductor longus and brevis. 10mL of local anesthetics were slowly injected. The needle was reinserted to position the needle tip on the fascia between adductor brevis and adductor magnus muscles, another 5mL of LA was injected.
  After that, the needle was reinserted to the same spots attached with nerve stimulator at 1.0 mA. If adductor muscle twitching was shown, another 5mL of LA was injected, and it was documented as 'fail'.
  nerve stimulator (stimuplex HNS12): whether using the nerve stimulator or not when the investigators do the ultrasound-guided obturator nerve block
  ultrasound: we did obturator nerve block with ultrasound guided method for searching the fascias where the anterior and posterior branches of obturator nerve run.
Arm/Group | US-IFI Group | US-NS Group
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31

LIMITATIONS AND CAVEATS:
We checked the success or fail with nerve stimulator only before beginning the surgery. Therefore, the possibility of incomplete anterior or posterior branch block due to the investigator's miss still remained, which is a limitation of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No